CLINICAL TRIAL: NCT03290157
Title: Evaluation of Improvement of Colonoscopy Preparation by Using a SPA
Brief Title: Improvement of Colonoscopy Preparation by Using a SPA
Acronym: ColoprAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Alexander Meining, Head of Endoscopy department, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ColoprAPP Study
Record Dates: First submitted 2017-09-15; First posted 2017-09-21 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Colonoscopy Preparation
Keywords: Colonoscopy; preparation; new media; SPA; APP

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Regular colonoscopy preparation paper based information provided
- ColoprAPP group (Other): Regular colonoscopy preparation paper based information provided plus usage of a downloaded SPA (ColoprAPP) as a reminder system for colonoscopy preparation
  Interventions: Device: ColoprAPP

INTERVENTIONS:
Device: ColoprAPP — Additional downloaded SPA for reminding the crucial steps of colonoscopy preparation
  Arms: ColoprAPP group

SUMMARY:
This study evaluates the impact of a SPA on Quality of bowel preparation for colonoscopy. Half of the patients receive regular paper based information on colonoscopy preparation (control), while the other half will use an additional SPA for colonoscopy preparation (coloprAPP).

DETAILED DESCRIPTION:
Preparation for colonoscopy is perceived as a major impediment to participate in CRC screening colonoscopy. Hence, inadequate bowel preparation is reported in up to 25% of all patients undergoing colonoscopy.

Although the quality of bowel preparation is influenced by various factors, it largely depends on patient´s compliance regarding instructions on purgatives and diet. Therefore reinforced education and guidance is a valuable tool to improve bowel preparation.

A rapidly increasing number of individuals worldwide use smartphones in their daily life. Application of this new technology into patient education could facilitate and empower the patient guidance. In this study patients either receive regular information on colonoscopy preparation (paper-based) or download a SPA for reinforced reminding of the steps of colonoscopy preparation. Objective of this study is to measure the impact of a SPA on quality of bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* smartphone
* outpatient appointment for colonoscopy
* CRC Screening, surveillance
* <ASA 3

Exclusion Criteria:

* no smartphone
* >ASA 3 (no possibility for outpatient colonoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-05-28 (Estimated)

PRIMARY OUTCOMES:
Quality of Bowel preparation | During colonoscopy procedure
  Measurement of bowel cleanliness by Boston Bowel preparation Scale (BBPS) with special regard on percentage of insufficient results of bowel preparation

SECONDARY OUTCOMES:
Adenoma detection rate | histological analysis after colonoscopy up to 10 days (d10)
  Rate of adenoma detected and resected during colonoscopy
Acceptance of patients towards bowel preparation procedure | at colonoscopy appointment (day 0)
  Measurement of patient satisfaction and acceptance with colonoscopy preparation procedure rated by numeric Rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Walter, MD, Principal Investigator — Universitätsklinikum Ulm
Locations (4):
- Germany (4):
  - Gastroenterologische Praxis Dornstadt, Dornstadt
  - Krankenhaus Landshut-Achdorf, Landshut
  - Krankenhaus Ludwigsburg, Ludwigsburg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Walter B, Frank R, Ludwig L, Dikopoulos N, Mayr M, Neu B, Mayer B, Hann A, Meier B, Caca K, Seufferlein T, Meining A. Smartphone Application to Reinforce Education Increases High-Quality Preparation for Colorectal Cancer Screening Colonoscopies in a Randomized Trial. Clin Gastroenterol Hepatol. 2021 Feb;19(2):331-338.e5. doi: 10.1016/j.cgh.2020.03.051. Epub 2020 Mar 30. PMID 32240835